CLINICAL TRIAL: NCT05510466
Title: Analysis of Efficiency and Tolerance of Triple BRAFinh/MEKinh /antiPD1 Combined Therapy in Patients With BRAF Mutated Melanoma With Central Nervous System Metastasis Occuring During First-line BRAFinh/MEKinh Therapy.
Brief Title: Triple BRAFinh/MEKinh /antiPD1 Combined Therapy in Patients With BRAF Mutated Melanoma With Central Nervous System Metastasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL22_0016
Record Dates: First submitted 2022-01-25; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-01

CONDITIONS: Metastatic Melanoma
Keywords: Initially treated by a doubled targeted therapy anti BRAF/anti MEK; immunotherapy; combined tritherapy; melanoma's brain metastasis; With an intra cerebral progression of the tumor
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Currently, therapeutic options in BRAF mutated melanoma with brain metastasis occurring after achievement of a good control of extracerebral secondary lesions by a first line combined targeted therapy (TT) are limited. In this setting, the addition of an anti PD1 agent to TT may be proposed as a second line strategy. This observational survey aims at investigating the benefit/risk ratio of this triple combination in a small cohort of patients.

ELIGIBILITY:
Inclusion criteria:

* Metastatic melanoma BRAF mutated
* Initially treated by a doubled targeted therapy anti BRAF/anti MEK
* With an intra cerebral progression of the tumor
* Whom we add an check point inhibitor anti PD1, combined with the double targeted therapy
* between 01/2019 et 01/2022

Exclusion criteria:

- Other condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Metastatic melanoma BRAF mutated
  * Initially treated by a doubled targeted therapy anti BRAF/anti MEK
  * With an intra cerebral progression of the tumor
  * Whom we add an check point inhibitor anti PD1, combined with the double targeted therapy
  * between 01/2019 et 01/2022
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-02-20 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
comparison between intra and extra cerebral metastasis | day 1
  comparison between intra and extra cerebral metastasis

CONTACTS AND LOCATIONS:
Overall Officials: Marie Louise Jeanne, resident, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC